CLINICAL TRIAL: NCT00685217
Title: Tension-free Vaginal Tape Management of Stress Incontinence in Women: Randomized Trial of TVT Secur Versus TVT
Brief Title: Transvaginal Tape (TVT) Secur Versus TVT Randomised Controlled Trial (RCT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other); Johnson & Johnson Medical Companies (Industry)
Responsible Party: Principal Investigator, Dr. Sue Ross, Adjunct Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21528
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TVT Secur surgical device (Experimental): Single incision tape device
  Interventions: Procedure: TVT Secur (Gynecare)
- TVT surgical device (Active Comparator): Usual care retropubic tape device
  Interventions: Procedure: TVT (Gynecare)

INTERVENTIONS:
Procedure: TVT Secur (Gynecare) — Sling device for stress urinary incontinence
  Arms: TVT Secur surgical device
Procedure: TVT (Gynecare) — Sling procedure for stress urinary incontinence
  Arms: TVT surgical device

SUMMARY:
This randomized multi-centre trial will recruit women with stress urinary incontinence who need surgical treatment for their condition. 300 women will be allocated either to receive a TVT Secur or a standard TVT surgical procedure. The main outcome is effectiveness of the procedure, determined using a 1-hour pad test (which tests for urine leakage) 12 months after surgery. The study will be carried out in 4 to 6 centers and will involve urogynaecologists, urologists and general obstetrician-gynaecologists: all clinicians will have received adequate training.

ELIGIBILITY:
Inclusion Criteria:

* Women with stress incontinence, defined as leaking with increased abdominal pressure
* Eligible for both types of surgery

Exclusion Criteria:

Women who:

* Have vaginal prolapse requiring surgical repair
* Have had previous incontinence surgery
* Have overactive bladder or incontinence is caused only by bladder overflow
* Intend to have further children
* Have Alzheimer's or Parkinson's disease, progressive neurological disease such as multiple sclerosis, or are immunocompromised
* Are unable to understand English
* Will be unavailable for follow-up

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Standardised pad test: "cure" is defined as less than 1g gain in pad weight over the duration of the test | 12 months following surgery

SECONDARY OUTCOMES:
Subjective evidence of cure | 12 months following surgery
Incontinence-related quality of life (UDI-6, IIQ-7) | 6 weeks and 12 months following surgery
Sexual function (PISQ-12) | 12 months following surgery
Satisfaction with surgical outcome | 12 months following surgery
  Patients will be asked about the expectations they had before surgery, and asked if the outcome had met expectations. Women will be asked about satisfaction with the surgical outcome, if they would have the same operation again under the same circumstances, and if they would recommend the same operation to someone else with the same problem.
Return to usual activities | up to 12 months following surgery
Voiding dysfunction | 12 months following surgery
Surgical complications | up to 12 months following surgery
Cost | up to 12 momths following surgery
Utility (15-D) | 6 weeks and 12 months following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sue Ross, PhD, Study Director — University of Calgary; Magali Robert, MD, Principal Investigator — University of Calgary; Jane Schulz, MD, Principal Investigator — University of Alberta
Locations (4):
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Penticton Regional Hospital, Penticton, British Columbia
  - Lions Gate Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share would depend on the protocol of an IPD analysis protocol

REFERENCES:
- [Result] Ross S, Tang S, Schulz J, Murphy M, Goncalves J, Kaye S, Dederer L, Robert M. Single incision device (TVT Secur) versus retropubic tension-free vaginal tape device (TVT) for the management of stress urinary incontinence in women: a randomized clinical trial. BMC Res Notes. 2014 Dec 22;7:941. doi: 10.1186/1756-0500-7-941. PMID 25532604